CLINICAL TRIAL: NCT02397928
Title: A Phase II Trial of Pemetrexed and Cisplatin or Carboplatin in Combination With TTFields (150 kHz) as First-line Treatment in Malignant Pleural Mesothelioma
Brief Title: Safety and Efficacy of TTFields (150 kHz) Concomitant With Pemetrexed and Cisplatin or Carboplatin in Malignant Pleural Mesothelioma (STELLAR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EF-23
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Malignant Pleural Mesothelioma; Treatment; Minimal toxicity; TTFields; Tumor Treating Fields; Novocure; Pemetrexed; Carboplatin; Cisplatin
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TTFields concomitant to pemetrexed plus cisplatin/carboplatin (Experimental): Patients will be treated continuously with TTFields, in addition to pemetrexed plus cisplatin/carboplatin
  Interventions: Device: NovoTTF-100L device; Drug: Pemetrexed; Drug: Cisplatin or Carboplatin

INTERVENTIONS:
Device: NovoTTF-100L device — Patients will be treated continuously with the NovoTTF-100L device. NovoTTF-100L treatment will consist of wearing four electrically insulated electrode arrays on the thorax. The treatment enables the patient to maintain regular daily routine.
  Other Names: TTFields
Drug: Pemetrexed — Pemetrexed 500 mg/m2 will be administered by intravenous infusion over 10 minutes or according to institutional administration timing on day 1 of a 21-day cycle.
Drug: Cisplatin or Carboplatin — Cisplatin 75 mg/m2 or carboplatin AUC 5 will be administered by infusion after adequate hydration according to institutional practices beginning approximately 30 minutes after the end on the pemetrexed infusion on day 1 of a 21-day cycle.

SUMMARY:
The study is a prospective, single arm, non-randomized, open label phase II trial, designed to study the safety and efficacy of a medical device, the NovoTTF-100L concomitant with Pemetrexed and cisplatin or carboplatin in Malignant Pleural Mesothelioma patients. The device is an experimental, portable, battery operated device for chronic administration of alternating electric fields (termed TTFields or TTF) to the region of the malignant tumor, by means of surface, insulated electrode arrays.

DETAILED DESCRIPTION:
PAST PRE CLINICAL AND CLINICAL EXPERIENCE:

The effect of TTFields has demonstrated significant activity in in vitro mesothelioma pre-clinical models both as a single modality treatment and in combination with pemetrexed and cisplatin, chemotherapies that are commonly used to treat malignant pleural mesothelioma.

In a pilot clinical trial (first in men) TTFields were shown to have an effect as a monotherapy in one patient with malignant pleural mesothelioma when applied to the patient's abdomen (the disease metastasized to the abdomen).

In a pilot study, 42 patients with stage IIIB- IV non-small cell lung cancer (NSCLC) who had had tumor progression after at least one line of prior chemotherapy received pemetrexed together with TTFields applied to the chest and upper abdomen until disease progression. Efficacy endpoints were remarkably high compared to historical data for pemetrexed alone.

In a large prospective, randomized trial, in recurrent glioblastoma (GBM). The outcome of subjects treated with TTFields was compared to those treated with an effective best standard of care chemotherapy (including bevacizumab). TTFields arm subjects had comparable overall survival to subjects receiving the best available chemotherapy in the US today. Similar results showing comparability of TTFields to best standard of care (BSC) chemotherapy were seen in all secondary endpoints. Recurrent GBM patients treated with TTFields in this trial experienced fewer side effects in general, significantly fewer treatment related side effects, and significantly lower gastrointestinal, hematological and infectious adverse events compared to controls. The only device-related adverse events seen were a mild to moderate skin irritation beneath the device electrodes. Finally, quality of life measures were better in TTFields Therapy subjects as a group when compared to subjects receiving effective best standard of care chemotherapy.

Recently, an interim analysis of a large ongoing phase III trial in newly diagnosed GBM showed that adding TTFields to the standard of care temozolomide chemotherapy significantly prolonged patients' progression free survival and overall survival. An independent data monitoring committee recommended to stop the trial for early success. The FDA approved cross over of control arm patients to the TTFields arm of the trial.

DESCRIPTION OF THE TRIAL:

All patients included in this trial are diagnosed with malignant pleural mesothelioma. In addition, all patients must meet all eligibility criteria.

Eligible patients will be enrolled, baseline tests will be performed and the patients will be treated continuously with the device concomitant with weekly pemetrexed and cisplatin or carboplatin until disease progression.

TTFields treatment will consist of wearing four electrically insulated electrode arrays on the thorax. Electrode array placement will require shaving of the chest/back as necessary before and during the treatment. After an initial short visit to the clinic for training and monitoring, patients will be released to continue treatment at home where they can maintain their regular daily routine.

During the trial the patient will need to return once every 3 weeks to the clinic where an examination by a physician and a routine laboratory examinations will be done. These routine visits will continue for as long as the patient's disease is not progressing. A routine CT scan of the chest and abdomen will be performed at baseline and every 6 weeks thereafter, until disease progression. After this follow up plan, patients will be contacted once per month by telephone to answer basic questions about their health status.

SCIENTIFIC BACKGROUND:

Electric fields exert forces on electric charges similar to the way a magnet exerts forces on metallic particles within a magnetic field. These forces cause movement and rotation of electrically charged biological building blocks, much like the alignment of metallic particles seen along the lines of force radiating outwards from a magnet.

Electric fields can also cause muscles to twitch and if strong enough may heat tissues. TTFields are alternating electric fields of low intensity. This means that they change their direction repetitively many times a second. Since they change direction very rapidly (150 thousand times a second), they do not cause muscles to twitch, nor do they have any effects on other electrically activated tissues in the body (brain, nerves and heart). Since the intensities of TTFields in the body are very low, they do not cause heating.

The breakthrough finding made by Novocure was that finely tuned alternating fields of very low intensity, now termed TTFields (Tumor Treating Fields), cause a significant slowing in the growth of cancer cells. Due to the unique geometric shape of cancer cells when they are multiplying, TTFields cause the building blocks of these cells to move and pile up in such a way that the cells physically explode. In addition, cancer cells also contain miniature building blocks which act as tiny motors in moving essential parts of the cells from place to place. TTFields cause these tiny motors to fall apart since they have a special type of electric charge.

As a result of these two effects, cancer tumor growth is slowed and can even reverse after continuous exposure to TTFields.

Other cells in the body (normal healthy tissues) are affected much less than cancer cells since they multiply at a much slower rate if at all. In addition TTFields can be directed to a certain part of the body, leaving sensitive areas out of their reach.

In conclusion, TTFields hold the promise of serving as a brand new cancer treatment with very few side effects and promising affectivity in slowing or reversing this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological or histological evidence of mesothelioma
2. ≥ 18 years of age
3. Not candidate for curative treatment (surgery or radiotherapy)
4. At least 4 weeks since major surgery
5. At least one measurable or evaluable lesion according to modified RECIST Criteria
6. ECOG Performance Status of 0-1
7. Life expectancy of at least 3 months
8. Participants of childbearing age must use effective contraception as indicated by the investigator
9. All subjects must sign written informed consent.
10. Able to operate the NovoTTF-100L System independently or with the help of a caregiver

Exclusion Criteria:

1. Patient candidate for surgery or radiotherapy with curative intent
2. Previous chemotherapy or radiation
3. Prior malignancy requiring anti-tumor treatment (apart from in-situ cervical cancer, in situ breast cancer, non-melanomatous skin cancers, or any malignancy for which treatment was received and there is no evidence of disease for at least 5 years) or concurrent malignancy
4. Significant co-morbidities within 4 weeks prior to enrollment, resulting in the following laboratory findings:

   1. Significant liver function impairment:

      * AST or ALT > 3 times the upper limit of normal
      * Total bilirubin ≥ 1.5 times upper limit of normal
   2. Significant renal impairment (serum creatinine > 1.7 mg/dL)
   3. Coagulopathy (as evidenced by PT or APTT >1.5 times control in subjects not undergoing anticoagulation)
   4. Thrombocytopenia (platelet count < 100 x 10^3/μL)
   5. Neutropenia (absolute neutrophil count < 1.5 x 10^3/μL)
   6. Anemia (Hb < 10 g/dL)
   7. Severe acute infection
5. Significant comorbidity which is expected to affect patient's prognosis or ability to receive the combined therapy:

   1. History of significant cardiovascular disease unless the disease is well controlled.

      Significant cardiac disease includes second/third degree heart block; significant ischemic heart disease; poorly controlled hypertension; congestive heart failure of the New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary activity results in fatigue, palpitation or dyspnea)
   2. History of arrhythmia that is symptomatic or requires treatment. Patients with atrial fibrillation or flutter controlled by medication are not excluded from participation in the trial
   3. Active infection or any serious underlying medical condition that would impair the ability of the patient to receive protocol therapy
   4. History of any psychiatric condition that might impair the patient's ability to understand or comply with the requirements of the study or to provide consent
6. Untreated brain metastases. Asymptomatic, pretreated brain metastases not requiring steroids are allowed
7. Implanted pacemaker, defibrillator or other electrical medical devices
8. Known allergies to medical adhesives or hydrogel
9. Pregnant or breast feeding (all patients of childbearing potential must use effective contraception method during the entire period of the study based on the recommendation of the investigator or a gynecologist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 1 year

SECONDARY OUTCOMES:
Progression Free Survival | 1 year
Response Rate | 1 year
Toxicity- incidence of adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Luca Ceresoli, MD, Principal Investigator — Cliniche Humanitas Gavazzeni
Locations (13):
- Antwerp University Hospital, Thoracic Oncology, Antwerp, Belgium
- Goustave Roussy - Cancer Campus Grand Paris, Villejuif, France
- Universitätsklinikum Halle (Saale), Halle, Germany
- Italy (5):
  - A.S.O. "SS Antonio e Biagio e Cesare Arrigo", Alessandria
  - Cliniche Humanitas Gavazzeni, Bergamo
  - Ospedale Villa Scassi, Genoa
  - Ospedaliera di Perugia, Perugia
  - Ospedaliero Universitaria Pisana, Pisa
- Erasmus Mc, Rotterdam, Netherlands
- Poland (3):
  - Medical University Gdansk, Gdansk
  - Katedra i Klinika Onkologii Uniwersytetu Medycznegi im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Klinika Nowotworów Pluca I Klatki Piersiowej, Warsaw
- Vall d' Hebron Institute of Oncology (VHIO) Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Pless M, Droege C, von Moos R, Salzberg M, Betticher D. A phase I/II trial of Tumor Treating Fields (TTFields) therapy in combination with pemetrexed for advanced non-small cell lung cancer. Lung Cancer. 2013 Sep;81(3):445-450. doi: 10.1016/j.lungcan.2013.06.025. Epub 2013 Jul 23. PMID 23891283
- [Background] Pless M, Weinberg U. Tumor treating fields: concept, evidence and future. Expert Opin Investig Drugs. 2011 Aug;20(8):1099-106. doi: 10.1517/13543784.2011.583236. Epub 2011 May 9. PMID 21548832
- [Background] Kirson ED, Giladi M, Gurvich Z, Itzhaki A, Mordechovich D, Schneiderman RS, Wasserman Y, Ryffel B, Goldsher D, Palti Y. Alternating electric fields (TTFields) inhibit metastatic spread of solid tumors to the lungs. Clin Exp Metastasis. 2009;26(7):633-40. doi: 10.1007/s10585-009-9262-y. Epub 2009 Apr 23. PMID 19387848
- [Derived] Ceresoli GL, Aerts JG, Dziadziuszko R, Ramlau R, Cedres S, van Meerbeeck JP, Mencoboni M, Planchard D, Chella A, Crino L, Krzakowski M, Russel J, Maconi A, Gianoncelli L, Grosso F. Tumour Treating Fields in combination with pemetrexed and cisplatin or carboplatin as first-line treatment for unresectable malignant pleural mesothelioma (STELLAR): a multicentre, single-arm phase 2 trial. Lancet Oncol. 2019 Dec;20(12):1702-1709. doi: 10.1016/S1470-2045(19)30532-7. Epub 2019 Oct 15. PMID 31628016